CLINICAL TRIAL: NCT05325801
Title: An Open-Label, Dose Finding Study to Investigate the Safety, Pharmacokinetics, and Preliminary Efficacy of BMCA and GPRC5D Dual Target CAR-T Cells Therapy in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of CAR-T Cells Targeting Both BCMA and GPRC5D in Treatment of Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, Prof., Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sirius
Record Dates: First submitted 2022-03-15; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMCA and GPRC5D dual target CAR-T cells （OriC321） (Experimental)
  Interventions: Biological: BMCA and GPRC5D dual target CAR-T cells(OriC321)

INTERVENTIONS:
Biological: BMCA and GPRC5D dual target CAR-T cells(OriC321) — Patients will receive lymphodepleting chemotherapy followed by a single infusion of OriC321

SUMMARY:
An Open-Label, Dose Finding Study to Investigate the Safety, Pharmacokinetics, and Preliminary Efficacy of BMCA and GPRC5D dual target CAR-T cells therapy in Patients with relapsed or refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated, written informed consent prior to any study specific procedures;
* Estimated life expectancy of minimum of 12 weeks;
* ECOG 0-2;
* Diagnosed as multiple myeloma according to the IMWG criteria;
* Evidence of cell membrane GPRC5D and/or BCMA expression, as determined by a validated immunohistochemistry (IHC) or flow cytometry of tumor tissue; Subjects should have measurable disease. At least meet one of the following criteria:

  1. If IgG type MM, serum M protein ≥10g/L; if IgA, IgD, IgE or IgM type MM, serum M protein ≥5g/L;
  2. urine M protein level ≥0.2g(200mg/24h);
  3. light chain type MM, serum free light chain (sFLC) ≥ 100mg / L and K/ λ FLC ratio is abnormal;
  4. there are extramedullary lesions;
* Subjects have had at least 3 prior lines of therapy including chemotherapy based on proteasome inhibitors (PIs) and immunomodulatory agents (IMiDs);
* Adequate organ functions

Exclusion Criteria:

* Active smoldering multiple myeloma;
* Active plasma cell leukemia;
* With organ amyloidosis;
* Central nervous system (CNS) involvement;
* Pregnant or breastfeeding;
* Hepatitis B virus (HBV) surface antigen (HBsAg) or hepatitis B core antibody-positive and detectable HBV DNA in peripheral blood; Hepatitis C virus (HCV) antibody and hepatitis C virus RNA in peripheral blood; Human immunodeficiency virus (HIV) antibody
* Uncontrolled Hypertension hypertension defined as a blood pressure (BP) ≥150/95 mmHg; Symptomatic heart failure per New York Heart Association Classification Class II, III or IV), Mean resting corrected QT interval corrected by Fridericia's formula (QTcF) > 470 msec (female), 450 msec (male) obtained from ECG; Baseline left ventricular ejection fraction (LVEF) below institution's lower limit of normal (LLN) or <50%;
* Have a history of another primary malignancy within 5 years prior to starting study treatment. Exceptions here are as follows: the disease under study; adequately treated basal or squamous cell carcinoma of the skin; cancer of the cervix in situ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity AEs/SAEs | 2 years after CAR-T cell infusion

SECONDARY OUTCOMES:
Concentration of CAR-T cells | 2 years after CAR-T cell infusion
Objective response rate (ORR) | 2 years after CAR-T cell infusion
Progression-free survival (PFS) | 2 years after CAR-T cell infusion
Duration of response (DOR) | 2 years after CAR-T cell infusion
Overall survival (OS) | 2 years after CAR-T cell infusion
Percentage of Patients With Negative Minimal Residual Disease (MRD) | 2 years after CAR-T cell infusion